CLINICAL TRIAL: NCT01302106
Title: Phase II Study of Clofarabine in Combination With Low Dose Cytarabine for Untreated Patients With Poor Risk Myelodysplastic Syndromes
Brief Title: Study of Clofarabine in Combination With Low Dose Cytarabine to Treat Myelodysplastic Syndromes
Acronym: CLO2009AISSM05
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: For increased induction mortality in older patients due to specific combinations of drugs, other clinical factors such as patient age and comorbidities.
Sponsor: Fondazione Italiana Sindromi Mielodisplastiche-ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO2009AISSM05; EudraCT number 2009-012755-23
Record Dates: First submitted 2010-12-22; First posted 2011-02-23 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Clofarabine; Low Dose Cytarabine; Poor risk MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Clofarabine combined with low dose Ara-C
  Interventions: Drug: Clofarabine plus low dose Ara-C

INTERVENTIONS:
Drug: Clofarabine plus low dose Ara-C — Clofarabine 10 mg/m2 by a 1-hr i.v infusion, once daily, from day 1 to 5. Ara-C 10 mg/m2, subcutaneously, twice a day (q12 hrs), from day 1 to 15. Clofarabine will be given 4 hours before the 2nd dose of Ara-C.

SUMMARY:
This is an interventional, multicenter, open label, phase II study designed to evaluate the safety and efficacy of Clofarabine in combination with low dose Cytarabine in untreated patients with poor risk of Myelodisplastic Syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 55 to 80 years
* Written informed consent to participate in the clinical trial
* Morphologically confirmed diagnosis of MDS according to WHO classification, and IPSS INT-2 or high risk according to IPSS index
* ECOG performance status 0-2
* No previous chemotherapy
* Serum bilirubin ≤1.5 times upper limit of normal (ULN) (unless elevation is due primarily to elevated unconjugated hyperbilirubinemia secondary to Gilbert's syndrome or hemolysis, but not to liver dysfunction)
* AST and ALT ≤2.5 times ULN
* Alkaline phosphatase ≤2.5 times ULN
* Serum creatinine ≤ 1 mg/dl: if serum creatinine > 1.0 mg/dl, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine) -1.154 x age in years -0-023 x 0.742 (if patient is female) x 1.212 (if patient is black)
* HIV negative

Exclusion Criteria:

* Have had any other chemotherapy or any investigational therapy as a treatment for MDS. Patients who received chemotherapy for other cancers than MDS/AML can be enrolled, provided that at least 6 months elapsed from accomplishment of the last course of chemo.
* Have had a prior hematopoietic stem cell transplant for MDS
* Have an uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Have a psychiatric disorder that would interfere with consent, study participation, or follow-up.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart
* Have had any prior treatment with Clofarabine
* Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy with the following exceptions: a.)Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease -free duration, are eligible for this study if definitive treatment for the condition has been completed. b.)Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.
* Have prior positive test for the Human Immunodeficiency Virus (HIV), HCV, HBV.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To assess the remission rate according to the combination regimen | 19 months

SECONDARY OUTCOMES:
Duration of response and survival | 19 months
Time to transformation in AML | 19 months
To determine the relationship of cytogenetic abnormalities and response to treatment | 19 months
To determine the safety and tolerability of the combination regimen | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Felicetto Ferrara, MD, Study Chair — Division of Hematology and Stem Cell Transplantation Unit, Ospedale "A.Cardarelli", Napoli, Italy
Locations (21):
- Italy (21):
  - SC Ematologia-AO SS.Antonio e Biagio e Cesare Arrigo, Alessandria
  - Dipartimento Scienze Mediche e Chirurgiche-Ospedale di Torrette, Ancona
  - Ematologia con trapianto-AO Policlinico Bari, Bari
  - SC di Ematologia-Spedali Civili, Brescia
  - centro di ricerca e di formazione ad alta tecnologia nelle Scienze-Università Cattolica Campobasso, Campobasso
  - Ematologia e Trapianto di Midollo Osseo-Ospedale Ferrarotto Alessi, Catania
  - Dipartimento di medicina Interna-Università di genova, Genova
  - UO Ematologia Vito Fazzi, Lecce
  - SC Ematologia-Azienda Ospedaliero Papardo, Messina
  - UO Ematologia-Ospedale San gennaro-ASL1, Napoli
  - Divisione di Ematologia e Trapianto Cellule Staminali-Ospedale A.Cardelli, Napoli
  - Medicina interna II- Azienda Ospedaliera S.Luigi Gonzaga, Orbassano
  - Divisione di Ematologia-Ospedale Vincenzo Cervello, Palermo
  - Dipartimento di Ematologia-Ospedale Spirito Santo Pescara, Pescara
  - Divisione di Ematologia- Azienda Ospedaliera Pisana Ospedale "S.Chiara", Pisa
  - Divisione Ematologia- AO Bianchi Melacrino Morelli, Reggio Calabria
  - UO Ematologia e Trapianto Cellule Staminali, IRCCS, Centro di Riferimento Oncologico della Basilicata, Rionero in Vulture
  - Ematologia-Azienda Ospedaliera Sant'Andrea, Roma
  - Divisione di Ematologia, Centro Trapianto di cellule staminali-IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo
  - UO Ematologia 2-Ospedale San Giovanni Battista, Torino
  - Divisione di Ematologia-Ospedale Cardinale Panico, Tricase